CLINICAL TRIAL: NCT03316014
Title: Adverse Drug Reactions in Pediatrics: Experience of a Regional Pharmacovigilance Center
Acronym: Pediatry ADR
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2016Ao003
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Child With Adverse Drug Reactions
Keywords: Pediatry; Adverse drug reactions; Pharmacovigilance
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Adverse Drug Reaction Reporting Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adverse drug reaction: Children from 0 to 17 years inclusive with ADR notifications recorded in the French pharmaco-vigilance database by the Regional Pharmacovigilance Center of Champagne-Ardenne between 1 January 1985 and 31 December 2014
  Interventions: Other: Adverse drug reaction

INTERVENTIONS:
Other: Adverse drug reaction — description of the adverse drug reactions (ADR) and the drugs involved in pediatrics

SUMMARY:
Aim. - To describe the adverse drug reactions (ADR) and the drugs involved in pediatrics.

Methods. - An observational study on all ADR notifications recorded in the French pharmaco-vigilance database by the Regional Pharmacovigilance Center of Champagne-Ardenne between 1 January 1985 and 31 December 2014 involving children from 0 to 17 years inclusive was performed. For all notifications, we studied the patient and the ADR characteristics

DETAILED DESCRIPTION:
Pediatry aged under 18 years accounted for around 22% of the French general population.

Data regarding drug safety from clinical trials are insufficient in this population.

Aim. - To describe the adverse drug reactions (ADR) and the drugs involved in pediatrics.

Methods. - An observational study on all ADR notifications recorded in the French pharmaco-vigilance database by the Regional Pharmacovigilance Center of Champagne-Ardenne between 1 January 1985 and 31 December 2014 involving children from 0 to 17 years inclusive was performed. For all notifications, we studied the patient and the ADR characteristics.

ELIGIBILITY:
inclusion criteria:

* Children from 0 to 17 years inclusive
* Who presented an adverse drug reaction notified to the Regional Pharmacovigilance Center of Champagne-Ardenne

exclusion criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Children from 0 to 17 years inclusive who presented an adverse drug reaction notified to the Regional Pharmacovigilance Center of Champagne-Ardenne.
Sampling Method: Non-Probability Sample
Enrollment: 632 (Actual)
Dates: Start 1985-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the different type of ADR | 30 years

REFERENCES:
- [Background] Saint-Martin C, Kanagaratnam L, de Boissieu P, Azzouz B, Abou Taam M, Trenque T. [Adverse drug reactions in pediatrics: Experience of a regional pharmacovigilance center]. Therapie. 2016 Oct;71(5):467-473. doi: 10.1016/j.therap.2016.04.001. Epub 2016 Apr 11. French. PMID 27203165